CLINICAL TRIAL: NCT05260502
Title: The Relationship Between Brain Volume and Sensory Integration in Children and Adolescence With Attention Deficit Hyperactivity Disorder and Autistic Spectrum Disorder.
Brief Title: The Relationship Between Brain Volume and Sensory Integration in Autistic and Attention Deficit Hyperactivity Disorder.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Moheb, principal investigator, Assiut University
Other Study IDs: Trbbvas
Record Dates: First submitted 2022-02-02; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Sensory Integration Dysfunction
Keywords: sensory disintegration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Autistic children: magnetic resonance imaging brain for autistic children
- attention deficit hyperactivity disorder children: magnetic resonance imaging brain for attention deficit hyperactivity disorder children
- Normal children: magnetic resonance imaging brain for Normal children

SUMMARY:
The relationship between brain volume and sensory integration in children and adolescence with attention deficit hyperactivity disorder and autistic spectrum disorder; comparative study

DETAILED DESCRIPTION:
Detect pattern of sensory disintegration in autistic and attention deficit hyperactivity disorder children and adolescence. Also detect relationship between changes in brain and sensory disintegration in each group.

ELIGIBILITY:
Inclusion Criteria .Diagnosis of Autism spectrum disorders /ADHD verified and confirmed on a clinical basis.

. Willing of the parents or the caregivers to participate in the study.

Exclusion Criteria:

.Children with intelligence quotient below 70. .Children with history or current substance use. .Children with medical or other neurological conditions. .Children with history of preterm labour (as brain volume lower than term delivery).

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Both males and females were included. Age ranges from 6- 18 years.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
sensory disintegration in neurodevelopmental disorders | 2 years
  Estimate the prevalence of sensory disintegration problems among study groups and differentiate the pattern of sensory disintegration problems among study groups.

REFERENCES:
- [Background] Gourley L, Wind C, Henninger EM, Chinitz S. Sensory Processing Difficulties, Behavioral Problems, and Parental Stress in a Clinical Population of Young Children. J Child Fam Stud. 2013 Oct 1;22(7):912-921. doi: 10.1007/s10826-012-9650-9. PMID 24443636
- [Background] Al-Heizan MO, AlAbdulwahab SS, Kachanathu SJ, Natho M. Sensory processing dysfunction among Saudi children with and without autism. J Phys Ther Sci. 2015 May;27(5):1313-6. doi: 10.1589/jpts.27.1313. Epub 2015 May 26. PMID 26157208
- [Background] Schaaf RC, Lane AE. Toward a Best-Practice Protocol for Assessment of Sensory Features in ASD. J Autism Dev Disord. 2015 May;45(5):1380-95. doi: 10.1007/s10803-014-2299-z. PMID 25374136